CLINICAL TRIAL: NCT03842384
Title: iENDURE: Digital Health Intervention to Support Opioid Use Disorder Treatment
Brief Title: Digital Health Intervention to Support Opioid Use Disorder Treatment
Acronym: iENDURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K23DA046482 (NIH); K23DA046482 (NIH)
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2023-03

CONDITIONS: Opioid Use Disorder; Treatment Adherence
Keywords: Buprenorphine; Digital Health; Medication for Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iENDURE (Experimental): iENDURE involves two delivery modes: computer and text message. The intervention initially targets motivational processes in combination with introductory strategies for managing physical and emotional distress through a single, brief, computer-delivered session followed by eight weeks of theoretically-informed text messages intended to enhance motivation and promote distress tolerance (DT).
  Interventions: Behavioral: iENDURE
- Treatment-as-Usual (No Intervention): Participants in the TAU comparison control group will engage in buprenorphine treatment as determined by their clinical team. This could include medication evaluations, individual or group counseling, case management or peer recovery. TAU was selected as the comparison condition as it represents a robust and evidence-based approach to the treatment of OUD.

INTERVENTIONS:
Behavioral: iENDURE — The proposed intervention will initially target motivational processes in combination with introductory strategies for managing physical and emotional distress through a single, brief, computer-delivered session followed by eight weeks of theoretically-informed text messages intended to enhance motivation and promote distress tolerance.
  Arms: iENDURE

SUMMARY:
In prior studies, the investigative team developed a combined computer- and text message-delivered personalized-feedback intervention (iENDURE) designed to enhance motivation and improve tolerance of distress to support the early phase of buprenorphine treatment. Specific aims of this subsequent study include conducting a preliminary randomized controlled trial with 80 participants to examine the efficacy of iENDURE relative to Treatment-as-Usual (TAU).

DETAILED DESCRIPTION:
Medication for Opioid Use Disorder (MOUD), which includes the use of Methadone, Buprenorphine, or long-acting Naltrexone, is an evidence-based approach to the treatment of Opioid Use Disorder. Buprenorphine, a partial opioid agonist, has grown in popularity over the last decade because of its safety profile and flexible administration. Despite its advantages, nearly half of participants are unable to achieve stabilization, and many discontinue treatment or return to illicit opioid use. Given high rates of noncompliance and/or dropout, there have been recent calls to find innovative interventions to enhance motivation, adherence, and retention in MOUD. Distress tolerance (DT), the perceived or actual ability to handle aversive physical or emotional states, is a transdiagnostic vulnerability factor implicated in the development and maintenance of affective symptoms/disorders and substance use. Preliminary work suggests that targeting DT during treatment may improve outcomes, by promoting the ability to persist in goal directed activity (e.g., abstinence) even when experiencing distress. Accordingly, an intervention that cultivates motivation for abstinence above the reinforcing effects of opioids and teaches adaptive distress tolerance strategies may optimize the induction and stabilization phases of buprenorphine treatment to improve long-term recovery. Personalized-feedback interventions, such as decisional balance feedback evaluating the advantages/disadvantages of engaging in a certain behavior, represent a promising method to enhance engagement in buprenorphine treatment. Digital health interventions have the capability of reaching a variety of patient populations and are well-suited to offer support, skills training, and reminders during times of increased distress that occur in 'real-time' outside of structured treatment settings. The objective of this study is to test the preliminary efficacy of a combined computer- and text message-delivered intervention for adults initiating buprenorphine treatment for opioid use disorder.

Following consent procedures, all participants will complete a brief online survey and then be randomly assigned to receive either (a) iENDURE, a computer- and text message-delivered intervention, or (b) treatment-as-usual and no additional intervention. All participants, regardless of treatment group, will complete a second set of questionnaires following randomization. All participants will also be scheduled for follow-up assessments at 1-, 4-, 8- and 12-weeks. Participants assigned to treatment-as-usual will engage in care as determined by their treatment team. Participants randomized to the iENDURE group will also engage in routine clinical care, however, they will additionally complete a brief computer intervention introducing designed to enhance motivation through a decisional balance exercise and improve tolerance of distress through skills training. Information obtained in the computer intervention will be used to personalize the subsequent text message portion of the intervention. Participants will receive 8 weeks of personalized text messages that will a) remind of salient motivational factors, and b) provide recommendations for relevant distress tolerance skills. Finally, participants in the iENDURE treatment condition will be asked to complete a individual qualitative interview at the conclusion of the intervention to elicit feedback for further improvement and refinement of the iENDURE program.

ELIGIBILITY:
Inclusion Criteria:

* age 18+ years; current DSM-5 diagnosis of Opioid Use Disorder; current buprenorphine prescription; and access to cell phone with text message capability.

Exclusion Criteria:

* active suicidality and/or psychosis; not fluent in English; not having a phone data plan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Self-Reported Buprenorphine Adherence | Participants will be asked to report on daily use up to 1-, 4-, 8- and 12- week following medication induction.
  The Timeline Follow-Back will be used to collect self-report data on daily buprenorphine adherence. Adherence is recorded as either 0 (prescribed dose not taken) or 1 (prescribed dose taken). Buprenorphine adherence will be operationalized as the percentage of days positive for buprenorphine administration.
Self-Reported Illicit Substance Use | Participants will be asked to report on daily use up to 1-, 4-, 8- and 12- week following medication induction.
  The Timeline Follow-Back will be used to collect self-report data on daily illicit substance use. Illicit substance use will be recorded as either 0 (no illicit substance use) or 1 (illicit substance use). Illicit substance use will be operationalized as the percentage of days positive for drug use (separate by drug class).
Biochemically Verified Buprenorphine Adherence | Performed at 1-, 4-, 8- and 12- week following medication induction.
  Urine samples will be collected and tested to confirm adherence to buprenorphine. A 5 ng/mL urine buprenorphine cutoff will be indicative of compliance with buprenorphine treatment.
Biochemically Verified Illicit Substance Use | Performed at 1-, 4-, 8- and 12- week following medication induction.
  Urine samples will be collected and tested to confirm or deny use of other illicit substances.

SECONDARY OUTCOMES:
Readiness Ruler | 1-, 4-, 8-, and 12-weeks post medication induction.
  Brief assessment of a person's present motivational state relative to changing a specific behavior. In this study, the Readiness Ruler will assess participants' motivation to change use of illicit opioids. The ruler is based upon a likert scale ranging from 1 (Definitely NOT Ready to Change) to 10 (Definitely Ready to Change). Higher scores reflect greater motivation to change.
Confidence Scale | 1-, 4-, 8-, and 12-weeks post medication induction.
  This item assesses participant's confidence in meeting their recovery goals. Participants are prompted "Please indicate to what extent you feel confident in reaching your goals for treatment" and were expected to respond on a 11-point Likert scale, ranging from "0" = "I do not think I will reach my goals" and "10" = "I think I will definitely reach my goals". Higher score indicated greater levels of confidence in meeting goals.
Distress Tolerance Scale | 1-, 4-, 8-, and 12-weeks post medication induction.
  The Distress Tolerance Scale is a 15-item self-report measure in which respondents indicate, on a 5-point Likert-type scale (1 = strongly agree to 5 = strongly disagree), the extent to which they can experience and withstand distressing psychological states. Higher total scores reflect greater ability to tolerate distress. The total score is computed as a mean, with a possible range of 1-5.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten J Langdon, PhD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Langdon KJ, Ramsey S, Scherzer C, Carey K, Ranney ML, Rich J. Development of an integrated digital health intervention to promote engagement in and adherence to medication for opioid use disorder. Addict Sci Clin Pract. 2020 Apr 29;15(1):16. doi: 10.1186/s13722-020-00189-4. PMID 32349790